CLINICAL TRIAL: NCT01932047
Title: Patients Who Refractory Cancer Conqueror for Bio New Drug Development Translational Research Establishment - Establishment of Personalized Cell Library
Brief Title: Patients Who Refractory Cancer Conqueror for Bio New Drug Development Translational Research Establishment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Do-hyun Nam, Principal Investigator, Samsung Medical Center
Other Study IDs: 2010-04-004
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Refractory Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — * The problem with the existing pre-clinical testing technology
    1. Efficacy evaluation using existing cell lines
    2. Existing preclinical animal models (The tumors produced by the cancer cells subcutaneously injected into immunodeficient mice)
  * The solution plan
    1. The development of patient-specific personalized cell library
    2. The development of stereotactic(orthotopic) personalized animal models with the patient-derived cell lines derived from patients
Oversight: Data Monitoring Committee: No

SUMMARY:
■ Unmet medical needs for Refractory cancer Conquest

- Many advanced cancers are still detected Despite remarkable technological advances for the early diagnosis of cancer in the field last 20 years.

In the type of progressive carcinoma is very high malignancy despite a variety of therapeutic target treatment for refractory cancer.

The refractory cancer patients who main focus of this research defined as the adult solid tumor patients who have failed standard therapy according to the criteria

NCCN / ASCO (American Society of imsangam) / KCSG (Study Group for chemotherapy).

The survival rate of refractory cancer patients are estimated to be 30-40% of the total patients with metastatic solid tumors and these refractory cancers are

difficult to deal with or control to conventional treatment so shows almost close to 100% mortality.

Therefore the new development of therapies for conquer of refractory cancer are urgently required.

■ Preclinical translational research Unmet Needs of Bio-new drug development for conquer of refractory cancer

- The stage of preclinical translational research (Translational Research) connects between the early stages of development and clinical trials in the stage drug development.

The establishment of foundation based on the translational research is very necessary and this must have proven ability to treat refractory cancer.

The most anti-cancer drugs developed by existing preclinical testing method actually does not show a remarkable effect in many cases in the clinical trials,

even if showed a remarkable inhibitory cancer effect in animal testing.

The exact molecular diagnosis to treat targets and paradigm for the development of new drugs at the same time requires for target treatment.

The tailored cell lines by patients and the proven technology by animal models and unmet need for preclinical translational research is increasing

DETAILED DESCRIPTION:
■ The specimen obtainer in surgery room contact with the manager of Institute Refractory Cancer Research team by calling to Medi-call system(Phone No.system T.9825).

The specimen obtainer gives the information of speciman to the manager .

The manager contact to the speciman deleverer and The speciman deleverer transported the specimens safely to the laboratory space.

The written informed consent form should obtained from the subject prior to the surgery.

In the case of blood samples, The total 15 ~ 20 ㎖ blood (only once) extracted from the subject and about 10 ~ 15 ㎖ blood is used for the genomic DNA extraction.

ELIGIBILITY:
Inclusion Criteria:

1. The patients who agreed and written consent to participate in this research
2. The patients who are scheduled for collection such as the patient tissue, pleural fluid, cerebro spinal fluid, blood samples for the purpose of surgery and diagnostics
3. The patients who diagnosed with cancer as below - GBM, Colon Cancer, Ovarian Cancer, Lung Cancer, Breast Cancer, Brain metastases, Lymphoma, Bone Metastatic Cancer , Gastric Cancer, Pancreatic Cancer, Gall bladder Cancer, Prostate Cancer, Kidney Cancer, Bladder cancer, Osteosarcoma, Soft tissue sarcoma, Head and neck cancer, 기타 Brain tumor

Exclusion Criteria:

* 1) Those who do not agree in writing to participate in research

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject diagnosed with cancer(GBM, Colon Cancer, Ovarian Cancer, Lung Cancer, Breast Cancer, Brain metastases, Bone Metastatic Cancer, Lymphoma, Gastric Cancer, Pancreatic Cancer, Gall bladder Cancer, Prostate Cancer, Kidney Cancer, Bladder cancer, Osteosarcoma, Soft tissue sarcoma, Head and neck cancer),and other Brain tumor
Sampling Method: Probability Sample
Enrollment: 1523 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-08 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
The amount of sample size | 10years
  ■ Target number of subjects (years) GBM : 120 case Colon Cancer : 200 case Gastric Cancer : 345 case Ovarian Cancer : 40 case Lung Cancer : 30 case Breast Cancer : 100 case Brain metastases : 120 case Bone metastases : 50 case Lymphoma : 10 case Pancreatic Cancer : 100 case Gall Bladder cancer : 20 case Prostate Cancer : 50 case Kidney Cancer : 100 case Bladder Cancer : 200 case Osteosarcoma : 15 case Soft tissue sarcoma : 50 case Head & neck cancer : 30 case Other Brain tumor : 100case
  - Total case : 1680 case

SECONDARY OUTCOMES:
The size of real tumor portion on obtained tumor specimen | 10 years
  1. In the samples of frozen tissue stored at -80 ° C are processed by the method Frozen Hematoxylin & Eosin Stain.
  2. The criteria of evaluation : tumor size, Tumor Area, Tumor Cell Density, Tumor Nucleus Amount, Necrosis.
  3. The Results are distincted by Accept, Intermediate, Fail.

OTHER OUTCOMES:
Genomic DNA Extraction from blood specimen | 10 years
  1. Using QIAGEN kit: QIAmp DNA mini kit (Cat. No. 51306)
  2. The Volume measurement: Using Spectrophotometer (Nanodrop, ND-1000)

CONTACTS AND LOCATIONS:
Overall Officials: Jueun Kim, Coordinator, Study Director — Institutional Refractory Cancer Research
Locations (1):
- Samsung Medical Center, Seoul, Gyunggido, South Korea